CLINICAL TRIAL: NCT01792778
Title: Post-Market Study Comparing the Clinical Performance Two Blood Control Safety Peripheral Intravenous Catheters: A Pilot Study
Brief Title: RIGHT IV Pilot Study
Acronym: RIGHT IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smiths Medical, ASD, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: RIGHT IV Pilot Study
Record Dates: First submitted 2013-02-08; First posted 2013-02-15 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Peripheral Intravenous Catheters
Keywords: IV Catheters; Blood control

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ViaValve Safety IV Catheter (Active Comparator): Catheter insertion using the ViaValve Safety IV Catheter.
  Interventions: Device: ViaValve Safety IV Catheter
- Insyte Autoguard BC [Blood Control] Shielded IV Catheter (Active Comparator): Catheter insertion using the Insyte Autoguard BC Shielded IV Catheter
  Interventions: Device: Insyte Autoguard BC [Blood Control] Shielded IV Catheter

INTERVENTIONS:
Device: ViaValve Safety IV Catheter — Insertion of the peripheral intravenous catheters into both upper extremities of subjects
  Arms: ViaValve Safety IV Catheter
Device: Insyte Autoguard BC [Blood Control] Shielded IV Catheter
  Arms: Insyte Autoguard BC [Blood Control] Shielded IV Catheter

SUMMARY:
The purpose of this pilot study is to collect the necessary information for determining the appropriate sample size of a statistically powered trial comparing the performance of two different blood control peripheral intravenous catheters.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Willing and able to independently sign an English Informed Consent
* Have adequate veins for placement of IV catheters in both right and left upper extremities

Exclusion Criteria:

* Currently taking anti-coagulation medication
* Have a known bloodborne disease or bleeding tendency
* Have a known fear or adverse reaction to needles or blood
* Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Clinical performance and acceptability | IV catheters will be inserted, secured to subjects, and then immediately removed. Data regarding the insertion process will then be immediately collected.
  Primary outcome measure will be a composite of user ratings evaluating clinical performance and acceptability of each device via a 6-point Likert questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Schwartz, MBA, MSN, RN, PHN, Principal Investigator — Smiths Medical
Locations (1):
- University of Minnesota Interprofessional Education and Resource Center, Minneapolis, Minnesota, United States